CLINICAL TRIAL: NCT03305939
Title: A Lifestyle Intervention Program for the Prevention of Type 2 Diabetes Mellitus Among South Asian Women With Prior Gestational Diabetes Mellitus.
Brief Title: Lifestyle Intervention IN Gestational Diabetes (LIVING)
Acronym: LIVING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); All India Institute of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIVING
Record Dates: First submitted 2017-06-21; First posted 2017-10-10 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Gestational Diabetes,Lifestyle,Type 2 DM
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized in to the intervention group will receive group sessions, monthly phone calls, and telephonic prompts (text/voice recording).
  Interventions: Behavioral: Life style Intervention
- Control (No Intervention): Control group participants will be referred to their usual doctor for ongoing management, with no attempt made to influence this. They will not get any part of the intervention but will receive the usual care (if any exists). Any abnormal OGTT results during the follow-up visits will be provided to the patient and their doctor. This is entirely consistent with current usual care.

INTERVENTIONS:
Behavioral: Life style Intervention — The intervention will include 4 face-to-face group sessions in the first 6 months, followed by remote support strategies and intensification counseling sessions when needed. Ongoing support and contact shown to be important in supporting behavior change will consist of reminders, and motivational messages for small actionable behaviors, delivered using mobile text or voice messages. Program intensification will be offered to women who fail to meet their weight goals by the 6 month time point. All phases of the program focus on self- management across 3 themes
  1. simple healthy eating and moderate physical activity messages;
  2. behavioral skills such as problem solving/goal setting/self-monitoring; and
  3. enhancing internal motivation, self-efficacy and self-management. The program is deliberately not prescriptive, and has a focus on sustainable behaviors and local context.
  Arms: Intervention

SUMMARY:
Investigators have taken the learning from various programs to develop a new lifestyle program (LIVING) that has a high probability of being feasible, acceptable and cost-effective in the South Asian context for women with prior Gestational Diabetes Mellitus (GDM). Investigators will optimize this intervention using an iterative, systems-based and user-centered approach. The intervention will be delivered by auxiliary nurse midwives or their equivalent in each participating hospital, representing a strategy of within-system task-shifting to augment scalability and sustainability. Investigators will then evaluate this in a Randomised Controlled Trial (RCT) to determine whether it will reduce the incidence of Type 2 Diabetes Mellitus (T2DM), in a manner that is affordable, acceptable and scalable. This project focuses on generating new knowledge around implementation of a preventive strategy embedded within existing health systems, using mixed-methods evaluation to inform on cost-effectiveness, acceptability and scalability. It represents a case study into "Integrated Innovation TM" incorporating a science component (a program based on behavior change theory that supports a multi-level approach to prevention by combining individually targeted strategies with social support), a social component (an innovative workforce strategy) and a sustainability component (a systems perspective for integration with existing health system infrastructure).

DETAILED DESCRIPTION:
Burden: Diabetes Mellitus is a major public health concern for both the developed and the developing countries. Globally 246 million people are affected with diabetes, and this will rise to 300 million by 2025. In India, around 25% of the 25 million pregnancies are associated with GDM, and this is increasing rapidly over time. Reported prevalence rates for GDM in Sri Lanka and Bangladesh are 13% and 10% respectively, although the Bangladesh estimate varied from 9.7% to 12.9% when different criteria were used.

Knowledge gap: There is knowledge gap on whether a resource- and culturally-appropriate lifestyle intervention program will be more effective and cost effective relative to usual care in delaying or preventing incidence of T2D among women in South Asia. Evidence from developed countries indicates that a low-intensity lifestyle intervention, integrated with antenatal care in the health system, optimizes healthy diet and attenuates physical activity decline in early pregnancy.

Study Design: An open-label parallel group pragmatic individual RCT with blinded primary endpoint adjudication will be performed. The RCT will be preceded by an intervention development and optimization phase.

Study Setting: This is an individual RCT in 1414 women from 24 hospitals (approx) in India (700 participants from 10-12 hospitals), Bangladesh (350 participants from 4 hospitals) and Sri Lanka (350 participants from 4 hospitals).

Sample Size: The inclusion of 1414 women with GDM from 24 hospitals (~60/hospital) will provide 90% power (2α=0.05) to detect a relative risk of ≤0.65, assuming that the control group cumulative incidence for change in glycaemic category will be at least 20% (median follow-up 24 months), and allowing for 20% drop out from trial (data) follow-up. A key secondary outcome is body weight; inclusion of 1414 women will provide 90% power to detect a difference of 1.8kg (assuming mean body weight of 64.2kg [sd 10.4]) in a control group.

The selection process of the respondents for the full scale trial: Study staff will recruit women with GDM at 24 to 34 weeks of gestation through a standard Oral Glucose tolerance test (OGTT) following International Association of the Diabetes and Pregnancy Study Groups (IADPSG) criteria. If a patient has undergone assessment of glycaemic status prior to 24 weeks' gestation, an OGTT is performed to confirm the diagnosis between 24 and 34 weeks' gestation, unless she is treated with an oral hypoglycaemic drug and/or insulin before 24 weeks, and satisfies the IADPSG criteria for diagnosis of GDM. If only Fasting Plasma Glucose (FPG) was done at 24-34 weeks, then the patient is categorized as GDM/overt diabetes/ normal on the basis of FPG value alone.

The inclusion criteria are the absence of T2DM (i.e. confirmation of Normal Glucose Tolerance (NGT), Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT)) at 3 to 18 months post-partum OGTT.

Program specific training: Site training will occur prior to enrollment of study participants. Training will be done either by the Central Coordinating Center (CCC) directly or through a trained member at the Regional Coordinating Center (RCC).Prior to finalizing the intervention, it will be optimized in a substantive formative phase in each participating country, to develop the training module and finalize the content and mode of intervention delivery. In each participating country, a barriers analysis through formative phase has been conducted to understand local contextual factors.

For stage 2: After 3 to 18 months of delivery childbirth, each individual respondent who consented at stage 1 to be contacted for participation in the study will be approached again for a post-partum OGTT. Those who will be diagnosed as Impaired Glucose Tolerance (IGT) or Impaired fasting Glucose (IFG) or with normal glycaemic status, and satisfy all inclusion criteria, will be enrolled in the study for the next 3 years. Those individuals diagnosed with T2DM will be excluded from the study and will be referred to the usual care of an endocrinologist.

Assignment of interventions: Allocation procedure (Randomization):

Participants will be recruited and then randomly allocated to intervention and control arms by central concealed randomization. Randomization will be conducted through a central, computer-based randomization service, and will be stratified by country; site and use of insulin during pregnancy.

Blinding: By necessity, neither site investigators nor participants will be blinded to allocation (intervention vs. usual care). However, all central study staff, statisticians and outcome adjudicators will remain blinded until final database lock.

Study arms: The intervention will include 4 face-to-face group sessions combined with remote on-going support, and an intensification offering when needed. However depending on outcomes during the optimization phase, the balance of face-to-face and remote contact might vary substantially overall and between countries. The intervention group will be linked up with the facilitator and will be followed up by the outcome assessor. Face-to-face sessions will be delivered by a trained facilitator using the existing Help-her training program optimized for each country. Eligible and consenting women will attend group sessions comprising not more than 10 women and will have baseline measures assessed prior to the commencement of the program. During session 1 the respondents will receive a program specific user manual and over the following weeks work through the behavioral skills sessions with the intervention facilitator. The participant manuals developed for the PregDiabCare pilot will undergo minor adaption for use in each country. Each session will last for 90 minutes. Following the face to face visits participants will also receive reminders and motivational messages related to small actionable behaviors delivered using mobile text /voice messages adapted from the World Health Organisation (WHO) Be He@lthy Be MOBILE manual.

In addition, at 26 weeks from the commencement of the intervention, women will undergo a review of progress. Program intensification will be offered to women who gain more than 2% of baseline weight (which accounts for transient weight fluctuations) will receive two intensification sessions of individualized coaching, and monthly phone coaching for the remaining 6 months, delivered by the trained facilitators. All phases of the program focus on self-management through small, feasible, and sustainable changes, by building knowledge and skills across 3 themes (1) simple healthy eating and moderate physical activity messages; 2) behavioral skills such as problem-solving / goal-setting / self-monitoring; and 3) enhancing internal motivation, self-efficacy, and self-management.

All participants will undergo six monthly follow up, including data collection by using specific case record forms (CRF) and blood sample collection to check the blood glucose level using HbA1c and OGTT at alternate 6 month follow up visits. If the HbA1c value is more than 6.5%, the participant is called for an OGTT. Participants who develop T2DM will not be followed up further. Participants who change glycaemic category but do not develop T2DM, as well as participants who continue in their glycaemic category, will be followed up.

Control group participants will be referred to their usual doctor for ongoing management, with no attempt made to influence this. Any abnormal OGTT results during follow up will be provided to the patient and their doctor. This is entirely consistent with current usual care.

Primary outcome: Proportion of women with change of glycaemic category, at or prior to final visit; from Normal Glucose Tolerance to Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT) or T2DM; or Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT) to Type 2 Diabetes Mellitus (T2DM).

Secondary outcomes: Mean change in fasting blood glucose, mean change in body weight ,mean change in waist circumference (cm), changes in mean systolic blood pressure (SBP),mean change in physical activity level , change in diet.

Data collection methods: Data will be collected at randomization and 6 monthly intervals thereafter, involving a brief case record form, with additional OGTT and HbA1c tests, alternately conducted at the follow up 6 monthly visits and both tests at the End of Study visit. Data will be captured electronically and data management will strictly comply with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) guidelines, utilizing Standard Operating Procedures established at participating institutes. Monitoring will be used to ensure quality and completeness of data, with an emphasis on central statistical monitoring to minimize costs.

Data Analysis plan: Analysis will be based on the principle of intention-to-treat. The effectiveness of the study intervention on the primary outcomes will be determined using Cox models for survival data, with censoring of participants who develop a subsequent pregnancy or type 2 DM during follow-up. Analyses of secondary outcomes will be conducted using standard statistical procedures applicable to dichotomous, categorical or continuous data as appropriate. However, any country level change detected during the analyses will be reported.

Research Ethics Approval: Ethics approval has been obtained from a number of ethics committees, including the University of Sydney Human Research Ethics Committee. In India, approvals from the Health Ministry Screening Committee and the All India Institute of Medical Sciences (Central Coordinating Centre) have been obtained as have approvals from each participating hospital. In Sri Lanka, approval has been obtained from the Ethics Review Committee, Faculty of Medicine, University of Kelaniya, which is accredited by the Ministry of Health. In Bangladesh, ethics committee approval from icddr,b has been obtained to allow involvement of all hospitals. The trial is registered with the Clinical Trials Registries of India and Sri Lanka.

Consent: Participants willing to take part in the study will be consented by trial centres using a two-stage consent process with written informed consent being obtained both at initial engagement during pregnancy, as well as prior to randomisation. Participants will be given adequate explanation about the study and will be given ample time to consider their trial participation. They will be given the opportunity to ask questions about the trial and what their participation involves, and will receive clarification from the investigator and other study staff. A written informed consent form (using appropriately translated versions where appropriate) will be signed and personally dated by the subject or by the subject's legally acceptable representative, and by the person who conducted the informed consent discussion. If a subject is unable to read or if a legally acceptable representative is unable to read, an impartial witness should be present during the entire informed consent discussion and must attest the written informed consent form. A copy of the signed written informed consent form will be given to the trial participant.

Donor: The study is funded under Global Alliance for Chronic Diseases (GACD) Grant (APP1093171) by National Health and Medical Research Council of Australia (NHMRC) and Indian Council of Medical Research (ICMR) GACD Grant.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be the absence of T2DM (i.e. confirmation of NGT, IFG or IGT) at 3 to 18 months post-partum OGTT.

Exclusion Criteria:

* Exclusion criteria will be limited to:

Travel time to hospital more than 2 hours (unless individual circumstances will not impede hospital attendance for study visits), lack of access to a mobile telephone, use of steroids during pregnancy (other than for lung maturation of the baby), confirmed case of Type 2 Diabetes, likelihood of moving residence in the next 3 years, refused consent .

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be women
Enrollment: 1612 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of women with a change of glycaemic category, at or prior to final visit | 3 years
  From Normal Glucose Tolerance to Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT) or T2DM; or Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT) to Type 2 Diabetes Mellitus (T2DM).

SECONDARY OUTCOMES:
Changes in fasting blood glucose as assessed by OGTT | 3 years
  Mean Change in fasting blood glucose status during the study period among the respondents
Change in body weight as assessed by the standard study weighing scale | 3 years
  Mean change in body weight during the study period among the respondents.
Change in waist circumference (in cm) as assessed by the standard study measuring tape | 3 years
  Mean change in waist circumference (in cm) during the study period among the respondents.
Change in systolic blood pressure (SBP) as assessed by Omron BP measuring machine | 3 years
  Changes in mean systolic blood pressure (SBP) during the study period among the respondents.
Change in physical activity level as assessed by Modified Global Physical Activity Questionnaire (MGPAQ) | 3 years
  Mean change in physical activity level during the study period among the respondents.
Change in dietary habits as assessed by Intake 24 (a 24-hour recall questionnaire) | 3 years
  Mean change in dietary practice during the study period among the respondents.

CONTACTS AND LOCATIONS:
Overall Officials: Anushka Patel, Ph.D, Principal Investigator — The George Institute; Nikhil Tandon, Ph.D., Principal Investigator — All India Institute of Medical Sciences
Locations (20):
- Bangladesh (4):
  - Marie Stopes Clinic, Dhaka
  - Azimpur Matenity Clinic, Dhaka
  - BIRDEM (Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders), Dhaka
  - Mohammadpur Fertility Services & Training Centre, Dhaka
- India (11):
  - M S Ramaiah Medical College, Bengaluru
  - PGIMER, Chandigarh
  - Madras Diabetes Research Centre, Chennai
  - Goa Medical College & Hospital, Goa
  - Fernandez Hospital Foundation, Hyderabad
  - King Edward Memorial (KEM) Hospital, Mumbai
  - TNM College & BYL Nair Ch.Hospital, Mumbai
  - Kalpavriksh Super Speciality Centre, New Delhi
  - JIPMER (Jawaharlal Institute of Postgraduate Medical Education and Research), Puducherry
  - Maharaja Agrasen Hospital, Punjābi Bāgh
  - Christian Medical College, Vellore
- Sri Lanka (5):
  - Castle Street Hospital for Women, Colombo
  - De Soyza Maternity Hospital, Colombo
  - Colombo South Teaching Hospital, Kalubowila
  - Negombo District General Hospital, Negombo
  - Colombo North Teaching Hospital, Ragama

IPD SHARING:
Plan to Share IPD: Yes
To be developed
Time Frame: To be determined
Access Criteria: To de determined

REFERENCES:
- [Background] Gupta Y, Kapoor D, Josyula LK, Praveen D, Naheed A, Desai AK, Pathmeswaran A, de Silva HA, Lombard CB, Shamsul Alam D, Prabhakaran D, Teede HJ, Billot L, Bhatla N, Joshi R, Zoungas S, Jan S, Patel A, Tandon N. A lifestyle intervention programme for the prevention of Type 2 diabetes mellitus among South Asian women with gestational diabetes mellitus [LIVING study]: protocol for a randomized trial. Diabet Med. 2019 Feb;36(2):243-251. doi: 10.1111/dme.13850. Epub 2018 Nov 29. PMID 30368898
- [Background] Tewari A, Praveen D, Madhira P, Josyula LK, Joshi R, Kokku SB, Garg V, Rawal I, Chopra K, Chakma N, Ahmed S, Pathmeswaran A, Godamunne P, Lata AS, Sahay R, Patel T, Gupta Y, Tandon N, Naheed A, Patel A, Kapoor D. Feasibility of a Lifestyle Intervention Program for Prevention of Diabetes Among Women With Prior Gestational Diabetes Mellitus (LIVING Study) in South Asia: A Formative Research Study. Front Glob Womens Health. 2020 Nov 27;1:587607. doi: 10.3389/fgwh.2020.587607. eCollection 2020. PMID 34816163
- [Background] Shanthosh J, Kapoor D, Josyula LK, Patel A, Gupta Y, Tandon N, Jan S, Teede HJ, Desai A, Joshi R, Praveen D. Lifestyle InterVention IN Gestational diabetes (LIVING) in India, Bangladesh and Sri Lanka: protocol for process evaluation of a randomised controlled trial. BMJ Open. 2020 Dec 13;10(12):e037774. doi: 10.1136/bmjopen-2020-037774. PMID 33318108
- [Derived] Gupta Y, Kapoor D, Lakshmi JK, Praveen D, Santos JA, Billot L, Naheed A, de Silva HA, Gupta I, Farzana N, John R, Ajanthan S, Bhatla N, Desai A, Pathmeswaran A, Prabhakaran D, Teede H, Zoungas S, Patel A, Tandon N; LIVING Collaborative Group. The incidence and risk factors of postpartum diabetes in women from Bangladesh, India and Sri Lanka (South Asia) with prior gestational diabetes mellitus: Results from the LIVING study. Diabetes Res Clin Pract. 2023 Oct;204:110893. doi: 10.1016/j.diabres.2023.110893. Epub 2023 Aug 31. PMID 37657646
- [Derived] Tandon N, Gupta Y, Kapoor D, Lakshmi JK, Praveen D, Bhattacharya A, Billot L, Naheed A, de Silva A, Gupta I, Farzana N, John R, Ajanthan S, Divakar H, Bhatla N, Desai A, Pathmeswaran A, Prabhakaran D, Joshi R, Jan S, Teede H, Zoungas S, Patel A; LIVING Collaborative Group. Effects of a Lifestyle Intervention to Prevent Deterioration in Glycemic Status Among South Asian Women With Recent Gestational Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e220773. doi: 10.1001/jamanetworkopen.2022.0773. PMID 35234881